CLINICAL TRIAL: NCT07151495
Title: The Additive Prognostic Value of Speckle Tracking Echocardiography Compared to Bernard's Staging in Patients Undergoing Mitral Valve Surgery
Brief Title: Additive Prognostic Value of PALS Compared to Bernard's Staging in Patients Undergoing MV Surgery
Acronym: PROSPECT-MIT
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Siena (Other)
Responsible Party: Sponsor
Other Study IDs: 7837
Record Dates: First submitted 2025-08-12; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Speckle tracking and 2D echocardiography — The study will involve only the collection of data obtained from routine clinical procedures and a telephone follow-up. Preoperative echocardiographic data and pre-operative left atrial speckle tracking data will be retrieved

SUMMARY:
Mitral valve prolapse is the most common cause of mitral regurgitation requiring surgery in developed countries. While cardiac surgery is recommended for symptomatic patients, in accordance with the ESC guidelines on valvular heart disease, indications for intervention in asymptomatic patients are mainly based on two-dimensional echocardiographic criteria: the presence of left ventricular systolic dysfunction or dilatation (end-systolic diameter ≥ 40 mm and/or ejection fraction ≤ 60%); or, in patients with preserved left ventricular systolic function, the occurrence of atrial fibrillation secondary to valvular disease or pulmonary hypertension (systolic pulmonary artery pressure > 50 mmHg); finally, significant left atrial dilatation (indexed left atrial volume ≥ 60 ml/m² or diameter ≥ 55 mm) also represents an indication. Mitral valve repair is preferred over valve replacement with a prosthesis, as it is associated with lower intraoperative mortality, better long-term survival, and fewer valve-related complications. However, the cut-off values derived from conventional echocardiography and used as indicators for surgical intervention may reflect an already severe and irreversible structural and functional cardiac alteration. Moreover, they do not consider more advanced imaging techniques such as speckle tracking echocardiography, which is now widely used in clinical practice and allows for a quantitative assessment of myocardial function through the analysis of myocardial fiber shortening in the cardiac walls. Several studies have shown that preoperative peak left atrial longitudinal strain (PALS) has prognostic value in predicting postoperative clinical outcomes in patients undergoing surgery for primary mitral regurgitation, as well as in predicting left atrial reverse remodeling; this prognostic relevance has also been observed in asymptomatic patients and in cases of less than severe mitral regurgitation. Furthermore, Bernard et al. demonstrated the prognostic value of a staging system for extra-valvular cardiac damage, assessed using two-dimensional echocardiographic data, in asymptomatic patients with moderate or severe mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe primary mitral regurgitation treated with cardiac surgery
* Age > 18 years
* Signed informed consent form/Substitute declaration in place of the signed informed consent form in the case of deceased patients

Exclusion Criteria:

* Known coronary artery disease
* Infective endocarditis
* Functional mitral regurgitation
* Presence of additional left-sided valvular heart disease greater than mild
* History of prior cardiac surgery
* History of rheumatic valvular disease
* Pregnancy
* Absence of a signed informed consent form/Absence of the signed substitute declaration in the case of deceased patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe primary mitral regurgitation treated with cardiac surgery
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
All cause or cardiovascular mortality | 3 months
  To determine the additive prognostic value for the primary outcome (all cause or cardiovascular mortality) of left atrial speckle-tracking echocardiography (PALS) over Bernard's staging

SECONDARY OUTCOMES:
Composite endpoint: all cause or cardiovascular mortality, new onset of atrial fibrillation, hospitalization for cardiovascular cause (heart failure, acute coronary syndrome) | 3 months
  To determine the prognostic value for the composite endpoint of Bernard'staging and of PALS in our cohort of patients

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Pasquini, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS

IPD SHARING:
Plan to Share IPD: No